CLINICAL TRIAL: NCT05475717
Title: A Multicenter, Randomized, Open-label Phase II Clinical Trial Evaluating Alprostadil Liposomal Injection in the Prevention of Contrast-induced Acute Kidney Injury in Patients Undergoing Percutaneous Coronary Intervention
Brief Title: A Study to Explore the Efficacy of Alprostadil Liposomes Injection in the Prevention of CI-AKI
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Voluntarily suspended the trial due to strategic adjustments
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HF1307-004
Record Dates: First submitted 2022-07-20; First posted 2022-07-27 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2022-10

CONDITIONS: Contrast-induced Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 20 µg group (Experimental): Patients will receive alprostadil liposome injection at 20 µg once daily (QD) for 4 days (1 to 3 hours before surgery and 3 days after surgery).
  Interventions: Drug: Alprostadil liposome injection
- 40 µg group (Experimental): Patients will receive alprostadil liposome injection at 40 µg once daily (QD) for 4 days (1 to 3 hours before surgery and 3 days after surgery)
  Interventions: Drug: Alprostadil liposome injection
- 80 µg group (Experimental): Patients will receive alprostadil liposome injection at 80 µg once daily (QD) for 4 days (1 to 3 hours before surgery and 3 days after surgery)
  Interventions: Drug: Alprostadil liposome injection
- blank control group (No Intervention): Patients will receive only basic hydration therapy which the experimental groups will receive.

INTERVENTIONS:
Drug: Alprostadil liposome injection — Alprostadil liposome injection, iv drip, QD×4 days (1 to 3 hours before surgery and 3 days after surgery)
  Other Names: Alprostadil liposome
  Arms: 20 µg group; 40 µg group; 80 µg group

SUMMARY:
This is a multicenter, randomized, open-label phase II clinical trial to evaluate alprostadil liposomal injection in the prevention of contrast-induced acute kidney injury in patients undergoing percutaneous coronary intervention.

DETAILED DESCRIPTION:
The trial is a multicenter, randomized, open-label, two-stage study. The trial period includes a screening period (up to 14 days), a treatment period (4 days), and a safety follow-up period (7 days ± 3 days). At least 368 patients with pre-PCI (percutaneous coronary intervention) are expected to be included, and all patients will be contrasted with non-ionic hypotonic/isotonic contrast media.

The trail will be divided into two stages. Three dose groups are set in the first stage: 20 µg/day, 40 µg/day and 80 µg/day. In the first stage, on the basis of hydration prevention, patients will randomized to receive 20, 40 or 80 µg/day of alprostadil liposome injection for 4 days (1 to 3 hours before surgery and 3 days after surgery), once a day. The blank control group will only receive hydration prophylaxis. In the second stage, according to the comprehensive evaluation of the data in the first stage, a dose group will be selected to continue to be enrolled. The primary outcome measure is the incidence of contrast-induced acute kidney injury within 72 hours after PCI. During the administration of alprostadil liposomal injection, vital signs, physical examination, ECOG performance status, laboratory test, ECG, adverse events and PK parameters will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to participate in this clinical trial and sign the informed consent voluntarily; 2.18≤age≤80 years old, gender is not limited; 3.Suffering from coronary artery disease and preparing to undergo elective PCI; 4.Serum creatinine>1.5 mg/dL or 30≤eGFR<60 mL/(min·1.73m^2), and meet at least one of the following risk factors:

1. Cardiac function class NYHA class III;
2. Age > 75 years old;
3. Anemia (baseline hematocrit: <36% in women, <39% in men);
4. Diabetes.

Exclusion Criteria:

1. Pre-perform emergency PCI;
2. Previously allergic to alprostadil similar products and contrast agents; used alprostadil within 3 days before the first administration;
3. Severe renal insufficiency: renal replacement therapy may be performed in a short period of time or eGFR<30 mL/(min·1.73m^2);
4. Severe heart failure (LVEF <35% or NYHA class IV), acute heart failure, and pulmonary edema;
5. Requires mechanical circulatory support therapy (intra-aortic balloon pump, catheter-based ventricular assist device, venous-arterial extracorporeal membrane oxygenation therapy, etc.);
6. Hypotension: systolic blood pressure < 90 mmHg;
7. Acute bleeding disorders or bleeding tendency, and the investigators believe that they are not suitable to participate in this trial;
8. Severe anemia (hemoglobin <60 g/L);
9. Active hepatitis B virus infection (positive hepatitis B virus surface antigen and the quantitative detection value of hepatitis B virus DNA exceeds the upper limit of the normal range of the research center), positive for any one of hepatitis C virus antibody, HIV antibody, and Treponema pallidum antibody;
10. Abnormal liver function (alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 3 times the upper limit of normal);
11. Contrast agents or known nephrotoxic drugs (aminoglycoside antibiotics, amphotericin B, vancomycin, antiviral drugs, non-steroidal anti-inflammatory drugs (except aspirin), Immunosuppressants, traditional Chinese medicines and proprietary Chinese medicines containing aristolochic acid, etc.) within 14 days before the first application of the test drug, or the use of drugs that protect the kidneys against AKI (N-acetylcysteine, sodium bicarbonate, aminophylline) within 3 days before the first application of the test drug;
12. Severe renal artery stenosis, and in the opinion of the the investigator, is unsuitable to participate in this trial;
13. Electrolyte disorders (serum potassium <2.5 mmol/L or serum sodium <125 mmol/L);
14. A history of glaucoma or ocular hypertension or gastric ulcer;
15. Interstitial pneumonia or mental illness or dementia;
16. Malignant tumors;
17. Have participated in drug clinical trials and used drugs within 3 months before screening;
18. Pregnant or breastfeeding, or patients who cannot use effective contraception during the study;
19. Other patients deemed unsuitable for participation in this trial by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2024-01-03 (Actual)

PRIMARY OUTCOMES:
Incidence of contrast-induced acute kidney injury within 72 hours after PCI | from baseline to 72 hours after PCI
  Incidence of contrast-induced acute kidney injury within 72 hours after PCI

SECONDARY OUTCOMES:
Changes in serum creatinine from baseline at 24 hours, 48 hours, and 72 hours after angiography | from baseline to 72 hours after angiography
  Changes in serum creatinine from baseline at 24 hours, 48 hours, and 72 hours after angiography
Changes in blood urea nitrogen from baseline at 24 hours, 48 hours, and 72 hours after angiography | from baseline to 72 hours after angiography
  Changes in blood urea nitrogen from baseline at 24 hours, 48 hours, and 72 hours after angiography
Changes in cystatin C from baseline at 24 hours, 48 hours, and 72 hours after angiography | from baseline to 72 hours after angiography
  Changes in cystatin C from baseline at 24 hours, 48 hours, and 72 hours after angiography
Changes in hs-CRP from baseline at 24 hours, 48 hours, and 72 hours after angiography | from baseline to 72 hours after angiography
  Changes in hs-CRP from baseline at 24 hours, 48 hours, and 72 hours after angiography
Changes in IL-6 from baseline at 24 hours, 48 hours, and 72 hours after angiography | from baseline to 72 hours after angiography
  Changes in IL-6 from baseline at 24 hours, 48 hours, and 72 hours after angiography
Incidence of renal replacement therapy after angiography during the study period | from baseline to 7 days after last dose
  Incidence of renal replacement therapy after angiography during the study
Adverse events | from baseline to 7 days after last dose
  Adverse events from baseline to 7 days after last dose, including symptoms, Abnormal laboratory test
Incidence of major adverse cardiovascular events (MACE) during the study period (recurrent angina, nonfatal myocardial infarction, acute heart failure, ventricular fibrillation, cardiac death) | from baseline to 7 days after last dose
  Incidence of major adverse cardiovascular events (MACE) during the study period (recurrent angina, nonfatal myocardial infarction, acute heart failure, ventricular fibrillation, cardiac death)

CONTACTS AND LOCATIONS:
Overall Officials: Wen Xu, Derector, Study Director — CSPC ZhongQi Pharmaceutical Technology Co., Ltd.
Locations (1):
- Beijing University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No